CLINICAL TRIAL: NCT03066713
Title: Post-prandial Glucose Response From Phytochemical Rich Potato Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Mattes, Principle Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 055-046
Record Dates: First submitted 2017-02-21; First posted 2017-02-28 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Glycemic Response; Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: A (Experimental): Skin On French Fry - breakfast Skin On French Fry - lunch Mashed Potatoes - dinner
  Interventions: Other: Skin On French Fry
- Experimental: B (Experimental): Skin Off French Fry - breakfast Skin Off French Fry - lunch Mashed Potatoes - dinner
  Interventions: Other: Skin Off French Fry
- Experimental: C (Experimental): Hash brown - breakfast Hash brown - lunch Mashed Potato - dinner
  Interventions: Other: Hash brown
- Experimental: D (Experimental): Pancake - breakfast Pretzels - lunch Macaroni - dinner
  Interventions: Other: Carbohydrate control

INTERVENTIONS:
Other: Skin Off French Fry — Skin Off French Fries will be provided at breakfast and lunch
  Arms: Experimental: B
Other: Skin On French Fry — Skin On French Fries will be provided at breakfast and lunch
  Arms: Experimental: A
Other: Hash brown — Hash brown potatoes will be provided at breakfast and lunch.
  Arms: Experimental: C
Other: Carbohydrate control — A pancake will be provided at breakfast, and pretzels will be provided at lunch.
  Arms: Experimental: D

SUMMARY:
Assess the impact of high antioxidant potato products on postprandial glycemic response and subsequent appetite and food intake.

DETAILED DESCRIPTION:
Preliminary results from anthocyanin rich potato products suggest that a reduced postprandial glycemic response might be expected from certain types of potato products and that phenolic antioxidants may play a critical role in predicting the physiological response from potato products. Further, if consumed early in the day, such as at breakfast, a reduced glycemic response may serve to mitigate appetite and food consumption later in the day. Investigators aim to better understand how characteristics of commercial potato products (i.e. frozen potato products) with different phenolic profiles and content, may alter postprandial glycemic response and subsequent appetitive behavior. Specifically, investigators will assess the glycemic response from a serving of potato products in the morning using continuous glucose monitoring. Further, appetite and subsequent food consumption later in the day will be assessed through appetite logs and continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-25, male or female

Exclusion Criteria:

* BMI outside 18.5-25

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Blood Glucose over 24 hours | 24 hours
  Samples taken every 5 minutes for 24 hours by a continuous glucose monitor

SECONDARY OUTCOMES:
Appetite | Every hour for 24 hours
  Questionnaire on hunger, fullness, desire to eat, prospective consumption, thirst taken hourly on the same day as the feeding intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided